CLINICAL TRIAL: NCT05299437
Title: Personalized Therapy of Metastatic Thyroid Cancer: Biological Characterization and Optimization With 124I PET Dosimetry
Brief Title: Metastatic Thyroid Cancer Therapy Optimization With 124I PET Dosimetry
Acronym: 131THEROPT124
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Carlo Chiesa (Other)
Collaborators: Associazione Italiana per la Ricerca sul Cancro (Other)
Responsible Party: Sponsor-Investigator, Carlo Chiesa, Medical Physics Expert, Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Organization: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AIRC 21939
Record Dates: First submitted 2022-03-07; First posted 2022-03-29 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Metastatic Differentiated Thyroid Cancer
Keywords: Thyroid cancer, dosimetry, 124-I, therapy optimization
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Optimized therapy (Experimental): Patients with ascertained metastatic differentiated thyroid cancer will be studied with FDG PET, CT, and for genetic characterization. 100 MBq of 124-I are administered for blood and PET lesion dosimetry.
  According Jentzen et al, good efficacy (Tumour Control Probability > 80%) is obtained with absorbed dose higher than 80 Gy to soft tissue metastases, and > 650 Gy to bone metastases. These values ae pursued with the limit of 2 Gy to blood.
  Only soft tissue lesions will be considered as target for the calculation of the complete response rate.
  However, for ethical reasons, therapeutic activity will be chosen in order to be effective both on soft tissue and bone lesions. Patients with too low predicted lesion absorbed dose even administering the Maximum Tolerable Activity (2 Gy to blood) will exit the protocol to receive the standard of care.
  Interventions: Drug: Radioiodine optimized therapy

INTERVENTIONS:
Drug: Radioiodine optimized therapy — 124-I blood and lesion dosimetry will be used to optimize the 131-I therapeutic activity. Both 124-I and 131-I administration will be performed after hormon withdrawal.
  Primary tumour tissue and circulating miRNA will be analyzed to check the genetic status.

SUMMARY:
Failure of conventional radioiodine therapy of metastatic differentiated thyroid cancer could be explained by:

* a suboptimal therapeutic approach, based on the administration of empirically fixed amount of radioactivity
* the presence of lesions with impaired iodine uptake, due to the expression of specific mutations

The study aims to:

* optimize therapy with pre-treatment 124-I blood and lesion dosimetry
* collect genetic data to check if specific mutations and/or miRNA over-expression could be related to low iodine uptake or to radioresistance

DETAILED DESCRIPTION:
TRIAL DESIGN

This is a one-stage, phase II, single-arm, bi-centric study. Enrollment centres are the Istituto Nazionale Tumori in Milan, and the Sacro Cuore Don Calabria Hospital in Negrar, close to Verona. Both centres are located in North Italy. 124-I is produced by cyclotron in Negrar Radiopharmacy unit, while high-activity 131-I therapy will be delivered in Milan.

Patients with ascertained metastatic differentiated thyroid cancer are studied with FDG PET and CT. 124-I blood and lesion PET dosimetry is used to optimize the 131-I therapeutic activity. The same 124-I PET scans are repeated 6 months after therapy as response assessment. 124-I and 131-I administration are performed after hormon withdrawal.

Primary tumour tissue and circulating miRNA will be analyzed to check the genetical features.

According to 124-I dosimetric PET data published by Jentzen et al, good efficacy (Tumour Control Probability > 80%) is obtained with absorbed dose > 80 Gy to soft tissue metastases, and > 650 Gy to bone metastases. Seen this difference, only soft tissue lesions are considered as target for the calculation of the complete response rate.

However, for ethical reasons, therapeutic activity will be chosen in order to be effective both on soft tissue and bone lesions. Patients with too low predicted lesion absorbed dose even administering the Maximum Tolerable Activity (2 Gy to blood) will exit the protocol to receive the standard of care.

PRIMARY END-POINT

Evaluation of complete response (CR) rate on soft tissue metastases 6 months after treatment, or later. The best response will be considered.

SECONDARY END-POINTS

Assessment of:

* acute toxicity rate and severity
* the association among pre-treatment glucose metabolism, 124-I uptake and therapy response
* the association among genetic mutations (BRAF V600E, TERT promoter, others) on thyroid cancer tissue, pre- and post-treatment miRNA expression, pre- and post-treatment glucose metabolism, iodine uptake, and 131-I therapy response

SAMPLE SIZE AND POPULATION

By considering a complete response (CR) rate in patients of soft tissue metastases after fixed activity approach as published by Klubo-Gwiezdzinska et al and by assuming an increment of 15% in CR rate after dosimetry-based administration, 46 evaluable patients will be required to test the above hypotheses.

ELIGIBILITY:
Inclusion Criteria:

* Histo-pathological diagnosis of DTC
* At least one documented non surgically-curable soft-tissue metastasis previously untreated
* ECOG performance status = 0 - 1
* Life expectancy > 6 months
* Females of childbearing age must have negative serum pregnancy test prior to registration and agree to use birth control throughout the study and for 6 months after completion of therapy
* Preserved hematologic and renal function (hemoglobin > 10 g/dL; WBC > 3500/uL; neutrophils > 50%; PLT > 100000/uL; albumin ≥ 2.5 g/dL; creatinine ≤ 2 mg/dL)
* Signed informed consent

Exclusion Criteria:

* All lesions surgically resectable
* Minimal lymph nodal disease (diameter < 1 cm, up to 2 nodes)
* Patient with skeletal metastases only
* Lung diffuse miliary micro-metastases
* Ongoing pregnancy
* Breast-feeding (enrollment could be considered after suspension)
* Refusal of male and female patients to use an effective contraception method during the study and for 6 months after completion of protocol therapy
* Impossibility to undergo follow-up procedures
* Presence of medical, psychiatric or surgical condition, not adequately controlled by treatment, which would likely affect subjects' ability to complete the protocol
* Assumption of any anti-tumor therapy including chemotherapy, biological or investigational drug treatments
* Assumption of any myelotoxic drugs
* Previous or concomitant assumption of Amiodarone
* Any other oncologic disease that required treatment in the last 5 years.
* Participation in a clinical trial in which an investigational drug was administered within 30 days or 5 half-lives prior to the study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-05-12 (Actual); Primary Completion 2024-03-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Response | 6 months, repeated through study completion, an average of 2 year
  Evaluation of complete response (CR) rate on soft tissue metastases 6 months after treatment, or later. The best response will be considered.
  RECIST 1.1 Evaluation of the best response rate on soft tissue metastases

SECONDARY OUTCOMES:
Association between presence/absence of metastatic pre-treatment FDG uptake and response | 6 months, repeated through study completion, for an average of 2 year
  Statistical tests will be applied to test the significance of the association.
Association between the presence/absence of specific mutations in neoplastic thyroid tissue and response | 6 months, repeated through study completion, for an average of 2 year
  Statistical tests will be applied to test the significance of the association.
Association between circulating miRNA deregulation and response | 6 months, repeated through study completion, for an average of 2 years
  Statistical tests will be applied to test the significance of the association.
Progression Free Survival interval (PFS) [months] from the first iodine treatment. | every 6 months or more frequently, through study completion, for an average of 2 years
  PFS will be assessed according to the standard clinical practice
Overall Survival [months] from the first iodine treatment. | At the end of the study, an average of 2 years
  Survival status will be collected

OTHER OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Through study completion, an average of 2 years
  The frequece and the grade of sialoadenitis as well as the occurrence of xerostomia will be reported as adverse event, as well as hematological toxicity nadir.

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Chiesa, PhD, Principal Investigator — Nuclear Medicine, Fondazione IRCCS Istituto Nazionale Tumori
Locations (2):
- Italy (2):
  - Nuclear Medicine, Ospedale Sacro Cuore - Don Calabria, Negrar, Verona
  - Nuclear Medicine, Fondazione IRCCS Istituto Nazionale Tumori, Milan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Klubo-Gwiezdzinska J, Van Nostrand D, Atkins F, Burman K, Jonklaas J, Mete M, Wartofsky L. Efficacy of dosimetric versus empiric prescribed activity of 131I for therapy of differentiated thyroid cancer. J Clin Endocrinol Metab. 2011 Oct;96(10):3217-25. doi: 10.1210/jc.2011-0494. Epub 2011 Aug 17. PMID 21849530
- [Background] Nagarajah J, Janssen M, Hetkamp P, Jentzen W. Iodine Symporter Targeting with 124I/131I Theranostics. J Nucl Med. 2017 Sep;58(Suppl 2):34S-38S. doi: 10.2967/jnumed.116.186866. PMID 28864610
- [Background] Jentzen W, Verschure F, van Zon A, van de Kolk R, Wierts R, Schmitz J, Bockisch A, Binse I. 124I PET Assessment of Response of Bone Metastases to Initial Radioiodine Treatment of Differentiated Thyroid Cancer. J Nucl Med. 2016 Oct;57(10):1499-1504. doi: 10.2967/jnumed.115.170571. Epub 2016 May 19. PMID 27199362
- [Background] Jentzen W, Hoppenbrouwers J, van Leeuwen P, van der Velden D, van de Kolk R, Poeppel TD, Nagarajah J, Brandau W, Bockisch A, Rosenbaum-Krumme S. Assessment of lesion response in the initial radioiodine treatment of differentiated thyroid cancer using 124I PET imaging. J Nucl Med. 2014 Nov;55(11):1759-65. doi: 10.2967/jnumed.114.144089. Epub 2014 Oct 20. PMID 25332440